CLINICAL TRIAL: NCT06858631
Title: IMpact of a Program of AerobiC Physical Exercise and Nutritional Therapy, on Quality of Life and Glycometabolic Compensation in Patients Undergoing Pancreatectomy
Brief Title: IMPact of AerobiC Exercise in Addition to Nutritional Treatment on Quality of Life After Pancreatectomy
Acronym: IMPACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mezza Teresa, Dr., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6706
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Tumors; Diabetes; Malabsorption
Keywords: Pancreatectomy; Quality of Life; Physical Exercise
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus; Malabsorption Syndromes; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Performing Physical Exercise (Experimental): Subjects will perferm 30-minute net aerobic exercise sessions at moderate intensity (3-5 METS, 60%-70% of maximum heart rate) three times per week. Participants may choose from walking, cycling, or swimming, with the option to alternate activities to enhance adherence to the program. Each session will include 10 minutes of warm-up (gradual increase in intensity); 30 minutes of aerobic exercise and 10 minutes of cool-down (gradual reduction of intensity and optional stretching). Total weekly exercise duration will be 150 minutes.
  Interventions: Behavioral: Physical Aerobic Exercise
- Control (No Intervention): Subjects will undergo usual nutritional and endocrinological follow up after pancreatectomy. They will not perform any physical aerobic exercise.

INTERVENTIONS:
Behavioral: Physical Aerobic Exercise — 30-minute net aerobic exercise sessions at moderate intensity (3-5 METS, 60%-70% of maximum heart rate) three times per week. Walking, cycling, or swimming, with the option to alternate activities to enhance adherence to the program. Each session will include 10 minutes of warm-up (gradual increase in intensity); 30 minutes of aerobic exercise and 10 minutes of cool-down (gradual reduction of intensity and optional stretching). Total weekly exercise duration will be 150 minutes
  Other Names: Physical activity
  Arms: Performing Physical Exercise

SUMMARY:
The goal of this interventional study is to assess the impact of a 6-month unsupervised aerobic exercise program on the quality of life of patients undergoing partial or total pancreatectomy. The main question it aims to answer is:

Does an aerobic exercise program improve physical functioning and overall quality of life in post-pancreatectomy patients?

Eligible participants will be assigned to either an exercise group or a control group. Quality of life will be evaluated using standardized scoring scales, with a focus on physical functioning. Secondary outcomes include changes in metabolic parameters (glycemia, HbA1c, lipid profile), BMI, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female patients who have undergone partial or total pancreatectomy
* Age ≥18 and ≤80 years
* Ability to understand and complete questionnaires and willingness to participate in periodic assessments
* No symptoms suggestive of cardiovascular issues (e.g., angina, dyspnea, palpitations, syncope)
* No evidence of ischemic heart disease, cardiomyopathy, valvular heart disease, myocarditis, autoimmune diseases, infections, or fractures that would contraindicate moderate-intensity aerobic activity

Exclusion Criteria:

* Age >80 or <18 years
* Cardiovascular, musculoskeletal, rheumatologic, or neurocognitive disorders contraindicating aerobic exercise
* 10-year cardiovascular risk >20% without cardiological/sports medicine evaluation
* Diagnosis of unresectable tumor
* Presence of metastases
* Pregnancy or breastfeeding
* Ongoing chemotherapy and/or radiotherapy
* BMI ≥30
* BMI ≤18.5

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in quality of life | 12 months
  Identify changes in the quality-of-life score from the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 (v3). The EORTC QLQ-C30 (v3) evaluates health status through nine multi-item scales: Five functional scales (physical, role, cognitive, emotional, social); three symptom scales (fatigue, pain, nausea/vomiting); one global health status scale. Additionally, six single-item scales assess symptoms commonly associated with neoplastic disease and its treatment (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).

SECONDARY OUTCOMES:
Detect changes in physical symptomps with the pancreas-specific PAN26 questionnaire. | 12 months
  Assess possible changes in physical symptomps with the pancreas-specific PAN26 questionnaire. The PAN26 questionnaire consists of 26 four-level items, producing seven multi-item scale scores (each composed of two to four items) and nine single-item scores.
Assessing changes in muscle power between subjects ongoing nutritional plan versus subjects ongoing nutritional plan and physical exercise | 12 months
  The subjects will be using their dominant hand, applies as much grip pressure as possible on the dynamometer. The assistant will record the maximum reading (kg). The subjects will repeat the test 3 times and the highest recorded value will be recorded to assess the subject's performance.
Detect changes in body mass index during the follow-up. | 12 months
  At each follow-up visit, height (m) and weight (kg) will be recorded. BMI will then be measured as kg/m².

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katsourakis A, Vrabas I, Papanikolaou V, Apostolidis S, Chatzis I, Noussios G. The Role of Exercise in the Quality of Life in Patients After Pancreatectomy: A Prospective Randomized Controlled Trial. J Clin Med Res. 2019 Jan;11(1):65-71. doi: 10.14740/jocmr3675. Epub 2018 Dec 3. PMID 30627280
- [Background] Yeo TP, Burrell SA, Sauter PK, Kennedy EP, Lavu H, Leiby BE, Yeo CJ. A progressive postresection walking program significantly improves fatigue and health-related quality of life in pancreas and periampullary cancer patients. J Am Coll Surg. 2012 Apr;214(4):463-75; discussion 475-7. doi: 10.1016/j.jamcollsurg.2011.12.017. Epub 2012 Feb 7. PMID 22321518
- [Background] Duijts SF, Faber MM, Oldenburg HS, van Beurden M, Aaronson NK. Effectiveness of behavioral techniques and physical exercise on psychosocial functioning and health-related quality of life in breast cancer patients and survivors--a meta-analysis. Psychooncology. 2011 Feb;20(2):115-26. doi: 10.1002/pon.1728. PMID 20336645
- [Background] Sweegers MG, Altenburg TM, Chinapaw MJ, Kalter J, Verdonck-de Leeuw IM, Courneya KS, Newton RU, Aaronson NK, Jacobsen PB, Brug J, Buffart LM. Which exercise prescriptions improve quality of life and physical function in patients with cancer during and following treatment? A systematic review and meta-analysis of randomised controlled trials. Br J Sports Med. 2018 Apr;52(8):505-513. doi: 10.1136/bjsports-2017-097891. Epub 2017 Sep 27. PMID 28954800
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Rock CL, Thomson CA, Sullivan KR, Howe CL, Kushi LH, Caan BJ, Neuhouser ML, Bandera EV, Wang Y, Robien K, Basen-Engquist KM, Brown JC, Courneya KS, Crane TE, Garcia DO, Grant BL, Hamilton KK, Hartman SJ, Kenfield SA, Martinez ME, Meyerhardt JA, Nekhlyudov L, Overholser L, Patel AV, Pinto BM, Platek ME, Rees-Punia E, Spees CK, Gapstur SM, McCullough ML. American Cancer Society nutrition and physical activity guideline for cancer survivors. CA Cancer J Clin. 2022 May;72(3):230-262. doi: 10.3322/caac.21719. Epub 2022 Mar 16. PMID 35294043